CLINICAL TRIAL: NCT02430922
Title: EVOLUTION STUDY, a Physician-inititated Trial Investigating the Efficacy of the Self-Expanding iVolution Nitinol Stent for Treatment of Femoropopliteal Lesions
Brief Title: a Physician-inititated Trial Investigating the iVolution Nitinol Stent
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-150106
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- iVolution stent (Experimental): Patient's treated with the iVolution stent from iVascular for the treatment of femoropopliteal lesions.
  Interventions: Device: iVolution nitinol stent

INTERVENTIONS:
Device: iVolution nitinol stent

SUMMARY:
The objective of this clinical investigation is to evaluate the short-term (up to 12 months) outcome of treatment by means of the self-expanding iVolution nitinol stent in symptomatic (Rutherford 2-4) femoropopliteal arterial stenotic or occlusive lesions.

ELIGIBILITY:
Inclusion Criteria:

1. De novo lesion located in the femoropopliteal arteries suitable for endovascular treatment
2. Patient presenting with a score from 2 to 4 according to the Rutherford classification
3. Patient is willing and able to comply with specified follow-up evaluations at the predefined time intervals
4. Patient is >18 years old
5. Patient understands the nature of the procedure and provides written informed consent, prior to enrollment in the study
6. Prior to enrollment, the target lesion was crossed with standard guidewire manipulation One target lesion is located within the native SFA: distal point 3 cm above knee joint
7. The target lesion has angiographic evidence of stenosis or occlusion
8. Length of the target lesion is ≤ 15 cm by visual estimation
9. Target vessel diameter visually estimated is ≥4 mm and ≤7 mm
10. There is angiographic evidence of at least one vessel-runoff to the foot

Exclusion Criteria:

1. Presence of a stent in the target vessel that was placed during a previous procedure
2. Presence of an aortic thrombosis or significant common femoral ipsilateral stenosis
3. Previous bypass surgery in the same limb
4. Patients contraindicated for antiplatelet therapy, anticoagulants or thrombolytics
5. Patients who exhibit persistent acute intraluminal thrombus at the target lesion site
6. Perforation at the angioplasty site evidenced by extravasation of contrast medium
7. Patients with known hypersensitivity to nickel-titanium or other study device components
8. Patients with uncorrected bleeding disorders
9. Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding
10. Life expectancy of less than 12 months
11. Ipsilateral iliac artery treatment before target lesion treatment with a residual stenosis > 30%
12. Use of thrombectomy, atherectomy or laser devices during procedure
13. Any patient considered to be hemodynamically unstable at onset of procedure
14. Patient is currently participating in another investigational drug or device study that has not reached the primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Primary Patency at 12 months | 12 months
  freedom from >50% restenosis at 12 months as indicated by an independently verified duplex ultrasound peak systolic velocity ratio (PSVR) <2.5 in the target vessel with no reintervention

SECONDARY OUTCOMES:
Technical Success | Procedure
Primary Patency at 1 & 6 months | 1 & 6 months
Freedom from Target Lesion Revascularization (TLR) at 1, 6 and 12 months | at all follow-up visits
Clinical Success at 1, 6 and 12 months | at all follow-up visits
  Clinical success at follow-up is defined as an improvement of Rutherford classification at 1-, 6- & 12-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.
Serious adverse events until follow-up completions | 1,6,12 months and interem visits
  Any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — Flanders Medical Research Program
Locations (4):
- Belgium (4):
  - Imelda Hospital, Bonheiden, Antwerp
  - A.Z. Sint-Blasius, Dendermonde, East-Flanders
  - Heilig-Hart Ziekenhuis, Tienen, Flemish Brabant
  - OLV Aalst, Aalst, Oost-Vlaanderen

IPD SHARING:
Plan to Share IPD: Undecided